CLINICAL TRIAL: NCT04728633
Title: Chemoembolization of Uveal Melanoma Hepatic Metastases Using 300mg of BCNU Dissolved in Lipiodol® Followed by Gelfoam® Embolization
Brief Title: Transarterial Chemoembolization for the Treatment of Uveal Melanoma With Liver Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20P.1076; JT 15505 (Other: JeffTrial Number)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Malignant Neoplasm in the Liver; Metastatic Uveal Melanoma; Stage IV Choroidal and Ciliary Body Melanoma AJCC V8
MeSH Terms: conditions — Uveal Melanoma | interventions — Carmustine; Ethiodized Oil; Iodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (carmustine, ethiodized oil, gelatin sponge) (Experimental): Patients undergo TACE by receiving an infusion of carmustine dissolved in ethiodized oil and an injection of gelatin sponge. Treatment repeats Q4W for bilobar disease or Q7W for unilobar disease in the absence of disease progression or unacceptable toxicity or until maximum clinical benefit is obtained.
  Interventions: Drug: Carmustine; Drug: Ethiodized Oil; Procedure: Transarterial Chemoembolization; Other: Medical Device Usage and Evaluation

INTERVENTIONS:
Drug: Carmustine — Given via infusion
  Other Names: 1,3-Bis(2-chloroethyl)-1-nitrosourea; 1,3-Bis(beta-chloroethyl)-1-nitrosourea; BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; WR-139021; SRI 1720; SK 27702; Nitrumon; Nitrourean; N,N''-Bis(2-chloroethyl)-N-nitrosourea; FDA 0345; Carmustinum; Carmustin; steroid taper initiated on day of discharge
Drug: Ethiodized Oil — Given via infusion
  Other Names: Lipiodol; Iodized Oil; Ethiodol; ETHIODIZED OIL,; 8008-53-5
Procedure: Transarterial Chemoembolization — Undergo TACE
  Other Names: TACE
Other: Medical Device Usage and Evaluation — Given gelatin sponge via injection

SUMMARY:
This phase II trial studies the effect of transarterial chemoembolization in treating patients with uveal melanoma that has spread to the liver (liver metastases). Transarterial chemoembolization involves the injection of a blocking agent (gelatin sponge, ethiodized oil) and a chemotherapy agent (carmustine) directly into the artery in the liver to treat liver cancers. Chemotherapy drugs, such as carmustine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. transarterial chemoembolization with carmustine in combination with ethiodized oil and gelatin sponge may help cause the tumors in the liver to shrink or disappear.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine the efficacy (clinical response) in terms of disease control rate (DCR) (complete response [CR] + partial response [PR] + stable disease [SD]) with chemoembolization of hepatic metastases with 300 mg of carmustine (BCNU) in ethiodized oil in metastatic uveal melanoma patients.

SECONDARY OBJECTIVES:

To investigate overall survival (OS) and progression-free survival (PFS) in uveal melanoma patients with hepatic metastases.

To assess the toxicity of the above treatment regimen.

OUTLINE:

Patients undergo transarterial chemoembolization (TACE) by receiving an infusion of carmustine dissolved in ethiodized oil and an injection of gelatin sponge. Treatment repeats once every 4 weeks (Q4W) for bilobar disease or once every 7 weeks (Q7W) for unilobar disease in the absence of disease progression or unacceptable toxicity or until maximum clinical benefit is obtained.

Steroid taper will begin the day of patient discharge. After completion of study treatment, patients are followed up at 30 days, and then every 2 months for up to 2 years.

After 3 years from first treatment, follow-up scans may occur every 16-20 weeks and labs every other month.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic uveal melanoma in the liver
* Tumor burden < 75%. Patients must have at least one tumor measuring >= 10 mm in longest diameter by magnetic resonance imaging (MRI) or triphasic computed tomography (CT) (if MRI is not available or contraindicated)
* No prior transarterial catheter-directed therapies. Prior hepatic tumor ablation, hepatic radiation or liver resection will be permitted as long as growing measurable liver tumors exists. Prior systemic treatments are allowed as long as there are no outstanding toxicities greater than grade 1
* Willingness and ability to give informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Serum creatinine =< 2.0 mg/dl
* Bilirubin =< 2.0 mg/ml. Exceptions will be made for patients with diagnosed Gilbert's Syndrome. In this instance, a bilirubin level =< 3.0 mg/ml will be allowed for this patients with this syndrome
* Albumin >= 3.0 g/dl
* No ascites
* Granulocyte count >= 1500/m^3
* Platelet count >= 150,000/m^3

Exclusion Criteria:

* Less than 18 years of age
* Previous liver-directed treatments including immunoembolization, chemoembolization, radioembolization, hepatic arterial perfusion, or drug-eluting beads
* Presence of life-limiting extrahepatic metastasis that requires systemic treatment within 3 months. However, radiation treatment of extrahepatic metastases such as bone, lymph nodes or subcutaneous metastases will be permitted while the patient is on study. Zometa or X-Geva to treat bone metastases will also be permitted. Immune check-point inhibitors while on study will NOT be permitted
* Portal vein occlusion, or inadequate collateral portal venous flow, as determined by MRI
* Known active viral or autoimmune hepatitis requiring treatments with serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) equal or greater than 5 times normal
* Presence of uncontrolled hypertension or congestive heart failure, or acute myocardial infarction within 6 months of entry
* Presence of any other medical conditions that imply a survival of less than six months
* Uncontrolled severe bleeding tendency or active gastrointestinal (GI) bleeding due to varices or main portal vein occlusion. Abnormal coagulation test must be corrected prior to the procedure
* History of life-threatening allergic reaction to iodinated contrast or BCNU despite pre-treatment with steroids
* Pregnant and/or breastfeeding women
* Presence of known untreated brain metastases. If patients have had previous treatment for brain metastasis, an MRI or CT of the brain must confirm the stabilization of the brain metastasis for more than 4 weeks
* Biliary obstruction, biliary stent, or prior biliary surgery including sphincterotomy but excluding cholecystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Best response to treatment | After the completion of cycle 2 of chemoembolization (1 cycle = 4 or 7 weeks)
  Response to treatment
Disease control rate (DCR) including complete response + partial response + stable disease | Up to 2 years
  All estimates of rates (e.g., DCR) will be presented with corresponding confidence intervals. For DCR, the method of Atkinson and Brown will be used to allow for the two-stage design using the criteria adapted from the international criteria proposed by Response Evaluation Criteria in Solid Tumors 1.03.

SECONDARY OUTCOMES:
Time to progression | From the first chemoembolization to the time when progression of liver metastases is confirmed, assessed up to 2 years
  Will be estimated by the Kaplan-Meier method.
Overall survival | From the first chemoembolization until death, assessed up to 2 years
  Will be estimated by the Kaplan-Meier method. Date and cause of death will be recorded. The cause of death will be categorized as either cancer-related or cancer unrelated.

CONTACTS AND LOCATIONS:
Overall Officials: Carin Gonsalves, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson Univeristy, Philadelphia, Pennsylvania, United States